CLINICAL TRIAL: NCT00006578
Title: Evaluation of the Relationship Between Immunologic Recovery After Highly Active Antiretroviral Therapy and the Ability to Mobilize CD34+ Stem Cells Following G-CSF Administration
Brief Title: Evaluation of Specific Infection-Fighting Cells For Prediction of Immune Response to Anti-HIV and Immune-Boosting Medication
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG A5072; AACTG A5072; Substudy ACTG A5085s
Record Dates: First submitted 2000-12-01; First posted 2001-08-31 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Granulocyte Colony-Stimulating Factor; HIV Protease Inhibitors; Ritonavir; Lamivudine; Stem Cells; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Antigens, CD34; abacavir; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; abacavir; amprenavir; Lamivudine; Filgrastim

INTERVENTIONS:
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Lamivudine
Drug: Filgrastim

SUMMARY:
The purpose of this study is to see if the amount of stem cells (cells that can develop into many kinds of cells) in the blood before anti-HIV drugs are taken can predict if the immune system will become stronger after anti-HIV drugs are given and if anti-HIV drugs can restore stem cells.

HIV infection has been shown to cause stem cells not to function well. Granulocyte colony-stimulating factor (G-CSF), which causes stem cells to go from the bone marrow (tissues in the bones where blood cells are formed) into the bloodstream, could possibly help boost immunity after anti-HIV treatment. This study examines the effects of G-CSF in helping the immune system become stronger after beginning anti-HIV treatment.

DETAILED DESCRIPTION:
In HIV infection, a progressive decline and/or dysfunction of several cell types is seen. It is thought that stem cell dysfunction or destruction may contribute to the hematologic and immunologic perturbations characteristic of HIV infection and may possibly limit the extent of immunologic recovery following HAART. This study proposes to investigate whether stem cell function and reserves are important in determining the extent of immune reconstitution following HAART.

Patients are stratified according to CD4 count. On Day 0, patients receive a 7-day cycle of subcutaneous granulocyte colony-stimulating factor (G-CSF). Blood samples are collected regularly, and on Day 14 patients undergo real-time HIV-1 RNA determinations. On Day 28, or sooner if HIV RNA is at least 1 log above baseline on Day 14, HAART consisting of daily receipt of abacavir, lamivudine, amprenavir, and ritonavir is initiated and continues until Week 76. Patients who achieve viral suppression (below 400 copies/ml of plasma HIV-1 RNA) by Week 26 are eligible to receive a second 7-day cycle of G-CSF at Week 28 and, if viral suppression continues through Week 50, a third cycle of G-CSF at Week 52. Patients are followed every 8 weeks for changes in viral load. Additionally, patients are monitored at regular intervals for surrogate markers of immunologic recovery and, during each cycle of G-CSF, for measurements of stem cell mobilization. Patients may also volunteer for A5085s (Bone Marrow Aspirate Substudy) at participating sites.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years of age.
* Have HIV levels of at least 1,000 copies/ml within 28 days prior to study entry.
* Have a CD4 cell count of 500 cells/mm3 or less in the 28 days prior to study entry.
* Have not had anti-HIV therapy or have had no more than 2 weeks of prior anti-HIV therapy 90 days prior to study entry.
* Are a good candidate for anti-HIV therapy.
* Agree to abstinence or use a barrier method of birth control during the study and for 12 weeks afterward.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have ever had cancer.
* Have used G-CSF or GM-CSF within 180 days prior to study entry.
* Are allergic to E. coli products (such as insulin or human growth hormone).
* Abuse drugs or alcohol.
* Are receiving or have had, within 14 days prior to study entry, treatment for an opportunistic (AIDS-related) infection.
* Have a medical condition that would interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cara Wilson, Study Chair
Locations (5):
- United States (5):
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of North Carolina, Chapel Hill, North Carolina